CLINICAL TRIAL: NCT01080911
Title: 0.05 vs. 0.1 Milligram Spinal Morphine for Reducing Morphine Requirement After Vaginal Hysterectomy With/Without Anterior and Posterior Vaginoplasty
Brief Title: 0.05 mg Versus 0.1 mg Spinal Morphine for Reducing Morphine Requirement After Vaginal Hysterectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Sirilak Suksompong, Associate Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Si073/2010
Record Dates: First submitted 2010-03-03; First posted 2010-03-04 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Pain
Keywords: Spinal morphine; Vaginal hysterectomy
MeSH Terms: conditions — Pain | interventions — Morphine; Analgesics, Opioid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- spinal morphine 0.05 mg (Experimental): spinal morphine 0.05 mg plus 0.5% heavy marcaine 3.5 ml
  Interventions: Drug: Morphine
- spinal morphine 0.1 mg (Active Comparator): spinal morphine 0.1 mg plus 0.5% heavy marcaine 3.5 ml
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — spinal morphine 0.05 mg
  Other Names: opioid
  Arms: spinal morphine 0.05 mg
Drug: Morphine — spinal morphine 0.1 mg plus 0.5% heavy marcaine 3.5 ml
  Other Names: Opioid
  Arms: spinal morphine 0.1 mg

SUMMARY:
This study aims to compare the effect of spinal morphine between the dose 0.05 mg and 0.1 mg on the amount of morphine during the first 24 hours postoperative.

ELIGIBILITY:
Inclusion Criteria:

* Female ASA 1-3
* Undergoing vaginal hysterectomy with/without anterior and posterior vaginoplasty
* Can operate PCA device

Exclusion Criteria:

* History of allergy to the study drugs
* History of bleeding tendency
* History of infection at the back
* Patient refuse to have spinal anesthesia
* History of CAD or CVD

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
the amount of 24 hours morphine | 24 hour

CONTACTS AND LOCATIONS:
Overall Officials: Sirilak Suksompong, MD, Principal Investigator — Department of Anesthesiology, Faculty of Medicine, Siriraj Hospital, Mahidol University
Locations (1):
- Faculty of Medicine, Siriraj Hospital, mahidol University, Bangkok, Thailand